CLINICAL TRIAL: NCT04359329
Title: Phase II Clinical Trial of Estradiol to Reduce Severity of COVID19 Infection in COVID19+ and Presumptive COVID19+ Patients
Brief Title: Estrogen Patch for COVID-19 Symptoms
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Sharon Nachman (Other)
Responsible Party: Sponsor-Investigator, Sharon Nachman, Director of Pediatric Infectious Diseases, Stony Brook University
Organization: Stony Brook University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBU-EstrogenPatch-COVID19
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2020-04

CONDITIONS: COVID
MeSH Terms: interventions — Ortho Evra

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Experimental): Estradiol Patch
  Interventions: Drug: Estradiol patch
- Control (No Intervention): No intervention

INTERVENTIONS:
Drug: Estradiol patch — Participant receives estradiol 100 micrograms/day for 7 days through a patch applied on the skin
  Arms: Active

SUMMARY:
The purpose of this study is to find out if estrogen, a female sex hormone, given as a patch placed on skin of COVID19 positive or presumptive positive patients for 7 days can reduce the severity of COVID19 symptoms compared to regular care.

This study has two study groups. One group will receive the study drug, a single-use Climara 25cm2 estrogen patch. The other group will receive standard of care.

Participants will be asked questions about their symptoms for up 6 times in up to 45 days.

DETAILED DESCRIPTION:
As the COVID19 pandemic has spread, it has been observed that adult men of all ages and older women are at higher risk of developing serious complications from infection with the virus. Animal model studies of SARS suggest that the age and sex difference in COVID19 symptom severity may be due to protective and acute actions of the female sex hormone estrogen. Animal and human studies support immune modulating effects of estrogen that are acute acting in viral infections and wound repair processes that may reduce the damaging effects of the virus on the lung and symptom severity.

Our hypothesis is that a short 7 day course of estradiol delivered in a transdermal patch applied to the upper buttock in COVID19+ or presumptive positive patients will be safe and will reduce symptom severity in adult men and older women when given prior to intubation. COVID19+ and presumptive positive patients not requiring intubation will be enrolled to the study and randomized to receive an estrogen patch or standard of care. Patients will be followed up at day 1, 7, 14 and 28 for clinical symptoms and disease outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male ≥ 18 years of age or female ≥ 55 years of age
* Documentation of COVID19 positivity or the presence of one or more of the following new onset (<7 days) clinical features defining presumptive COVID19

  1. fever of >100.5°F or 38°C
  2. shortness of breath
  3. cough
  4. radiologic evidence of pneumonia
* Able to provide informed consent
* Able to be contacted by telephone for follow-up

Exclusion Criteria:

* Currently receiving estrogen based hormonal therapy
* Abnormal genital bleeding
* Protein C or Protein S deficiency
* Pre-existing liver impairment (e.g. Hepatitis C, cirrhosis)
* History of anaphylactic reaction or angioedema with Climara
* Receiving lamotrigine therapy
* Subjects with known past diagnosis of estrogen receptor positive breast cancer or endometrial cancer
* Subjects with severe hypoxia at risk for acute intubation in ED
* History of stroke
* Any history of thromboembolic event including deep vein thrombosis or pulmonary emboli
* Current use of St. John's Wort
* Males on testosterone
* History of myocardial infarction, cardiac stents, or active angina

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Rate of Hospitalization | 30 days
  Admission to hospital due to COVID-19 symptoms
Rate of Transfer to Intensive Care Unit | 30 days
  Occurrence of admission to ICU due to COVID-19 symptoms
Rate of Intubation | 30 days
  Occurrence of intubation
Rate of Death | 30 days
  Occurrence of death from COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Nachman, MD, Principal Investigator — Stony Brook University Hospital
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sultana J, Crisafulli S, Gabbay F, Lynn E, Shakir S, Trifiro G. Challenges for Drug Repurposing in the COVID-19 Pandemic Era. Front Pharmacol. 2020 Nov 6;11:588654. doi: 10.3389/fphar.2020.588654. eCollection 2020. PMID 33240091